CLINICAL TRIAL: NCT02349789
Title: Stimulating the Little Brain to Make Big Steps: Improving Gait in Parkinson's Disease Patients by Non-invasive Electrical Stimulation of the Cerebellum.
Brief Title: The Role of Cerebellar Hyperactivity in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other); University of Twente (Other)
Responsible Party: Principal Investigator, Amy J. Bastian, Ph.D., Ph.D., PT, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: IRB00052263
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease
Keywords: Gait; Cerebellum; Non invasive electrical stimulation; tDCS; TMS; Balance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Gait and balance disturbances are one of the most incapacitating symptoms of Parkinson's disease (PD) (Boonstra et al. 2008). They can cause falls and are therefore associated with the negative spiral of (near) falls, fear of falling, fractures, reduced mobility and social isolation; hence, having a profound negative impact on quality of life (Lin et al. 2012). Originally, symptoms of PD were ascribed to dopamine deficiency and basal ganglia dysfunction (Wu et al. 2013). However, in the last decades it has become clear that other brain structures are also involved in the pathophysiology of PD (Snijders et al. 2011; Stefani et al. 2007). An intriguing, emerging insight is that the cerebellum may be involved in the pathophysiology of PD (Wu et al. 2013). That is, the cerebellum is hyperactive in PD patients during different motor tasks (Yu et al. 2007; Hanakawa et al. 1999; del Olmo et al. 2006). However, whether cerebellar hyperactivity is pathological or compensatory and how it affects gait and balance in PD patients remain open questions. Here, the investigators aim to elucidate the role of the hyperactive cerebellum in gait dysfunction in PD patients by modulating cerebellar excitability with state-of-the-art non-invasive brain stimulation techniques and investigate the effects on gait.

DETAILED DESCRIPTION:
The cerebellum plays an important role in generating well-coordinated locomotion, voluntary limb movements and eye movements (Morton et al. 2004). It is particularly important for balance and limb coordination needed to generate a stable gait pattern (Morton et al. 2006). Specific roles of the cerebellum for gait include coordinating the two legs to produce a stable rhythmic pattern, dynamic regulation of balance, and adaptation of the pattern through practice (Morton et al. 2004). Though the core deficits of PD patients are largely different than those of cerebellar patients, they do show decreased bilateral coordination (Plotnik et al. 2008) and a fundamental disturbance in stride length regulation (Morris et al. 1998) during walking.

Recent work has shown that the cerebellum is hyperactive in PD patients, though it is not known whether this activity is compensatory (i.e. reduces motor impairments) or pathological (i.e. causes motor impairments). One idea is that increased cerebellar activity, affecting cerebral motor areas, compensates for the reduced drive from the basal ganglia (Wu et al. 2013). Alternatively, it is possible that cerebellar hyperactivity is pathological, as recent work suggests that cerebellar activity may be partially responsible for the generation of Parkinsonian tremor (Helmich et al. 2012). One approach to answer this question is to use non-invasive brain stimulation techniques to decrease the activity of the cerebellum in PD patients and determine if they improve or worsen their gait pattern.

Non-invasive brain stimulation techniques, such as transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS) are able to alter the excitability of brain pathways. Applying these techniques over the motor cortex, improved motor function in different patient groups, including stroke and PD (Benninger et al. 2010). Only two studies have investigated the effect of modulation of cerebellar-motor cortex excitability on motor function in PD patients. That is, 1 Hz repetitive TMS (inhibitory rTMS) over the cerebellum improved gross arm movements, but worsened fine motor skills17. Furthermore, a two-week continuous theta burst stimulation TMS protocol decreased levodopa-induced dyskinesias (Koch et al. 2009). These studies only investigated the effects on the upper extremities. The cerebellum is also hyperactive during gait (Hanakawa et al. 1999; del Olmo et al. 2006), but whether modulation of cerebellar excitability can improve gait deficits in PD patients is currently unknown.

Non-invasive brain stimulation can also be used to study the connection between the cerebellum and the motor cortex via using paired-pulse TMS. Specifically, cerebellar stimulation 5 ms before motor cortex stimulation leads to a reduction in the amplitude of motor-evoked potentials (MEPs), a phenomenon referred to as cerebellar-brain inhibition (CBI) (Pinto et al. 2001). This measure of CBI is abnormal in PD patients-it is reduced at rest, but increases with muscle contraction (Ni et al. 2010).

Gait impairments in PD are often resistant to treatment, particularly as the disease progresses. Therefore, insight in the pathophysiology of gait disturbances is essential for improving treatment options and quality of life for PD patients. This study will answer the question of whether cerebellar hyperactivity alleviates or worsens gait deficits in PD patients. If cerebellar hyperactivity in PD is compensatory, anodal (i.e. excitatory) tDCS should improve gait in PD patients, whereas cathodal (i.e. inhibitory) tDCS will make matters worse. In contrast, if cerebellar hyperactivity is pathological, cathodal tDCS will improve gait and anodal tDCS will worsen it. Hence, this study will improve the fundamental understanding of gait pathophysiology in PD patients. The investigators will focus on the aspects of gait that are particularly affected in PD and associated with fall risk, such as stride length and gait speed (Paul et al. 2013). In this way, this study may identify the cerebellum as a potential new target for treatment, opening up new possibilities improving gait and balance disturbances in PD.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate (Hoehn and Yahr scale: 1.5-3) idiopathic, akinetic-rigid type Parkinson's disease.
* Capable of walking for 5 minutes.

Exclusion Criteria:

* Severe dyskinesia
* Congestive heart failure.
* Peripheral artery disease with claudication.
* Cancer. Pulmonary or renal failure. Unstable angina. Uncontrolled hypertension (> 190/110 mmHg). Brain injury. History of seizure or a family history of epilepsy. Metal anywhere in the head except the mouth. Cardiac pacemakers. Cochlear implants. Implanted medication pump. Heart disease. Intracardiac lines. Increased intracranial pressure, such as after infarctions or trauma. Currently taking tricyclic anti-depressants or neuroleptic medication. History of head trauma. History of respiratory disease. Dementia (Montreal Cognitive Assessment < 26; Frontal Assessment Battery < 13). Orthopedic or pain conditions. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2017-09

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bastian, PT, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted by the following means: Subjects were referred by local physicians and recruited from databases of previous studies of Co-investigators. Flyers were disseminated locally.
Groups:
- Parkinson's Subjects: Participants with akinetic, rigid Parkinson's disease
Period: Overall Study
Arm/Group | Parkinson's Subjects
Started | 11
Completed | 9
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed- Sham_On
Description: Change in overground walking speed (10 meter walk test) after Sham transcranial direct current stimulation, participants on medication.
Time Frame: One session
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 9
meters per second (m/s) | -0.0185 (0.0255)

2. Primary Outcome: Change in Gait Speed- Sham_Off
Description: Change in overground walking speed (10 meter walk test) after Sham transcranial direct current stimulation, participants off medication.
Time Frame: One session
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 9
meters per second (m/s) | 0.0078 (0.01076)

3. Primary Outcome: Change in Gait Speed- Anodal_On
Description: Change in overground walking speed (10 meter walk test) after Anodal transcranial direct current stimulation, participants on medication.
Time Frame: One session
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 9
meters per second (m/s) | -0.0477 (0.01947)

4. Primary Outcome: Change in Gait Speed- Anodal_Off
Description: Change in overground walking speed (10 meter walk test) after Anodal transcranial direct current stimulation, participants off medication.
Time Frame: One session
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 9
meters per second (m/s) | 0.0346 (0.02359)

5. Primary Outcome: Change in Gait Speed- Cathodal_On
Description: Change in overground walking speed (10 meter walk test) after Cathodal transcranial direct current stimulation, participants on medication.
Time Frame: One session
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 9
meters per second (m/s) | -0.0059 (0.01908)

6. Primary Outcome: Change in Gait Speed- Cathodal_Off
Description: Change in overground walking speed (10 meter walk test) after cathodal transcranial direct current stimulation, participants off medication.
Time Frame: One session
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Parkinson's Subjects
Number analyzed (Participants) | 9
meters per second (m/s) | -0.0502 (0.02521)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months ( entire course of the study)
Arm/Group | Parkinson's Subjects
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT02349789/Prot_SAP_000.pdf